CLINICAL TRIAL: NCT03546127
Title: Molecular Profiling to Improve Outcome of Patients in Cancer. A Pilot Study (MULTIPLI-0)
Brief Title: Molecular Profiling to Improve Outcome of Patients in Cancer. A Pilot Study
Acronym: MULTIPLI-0
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Institut Bergonié (Other); Plateforme labellisée Inca - Institut Bergonié, Bordeaux (Unknown); Plateforme labellisée Inca - Hôpital Européen Georges Pompidou, Paris (Unknown); CNRGH, Evry (Unknown); EUCLID Clinical Trial Platform (Other)
Responsible Party: Sponsor
Other Study IDs: C17-11 MULTIPLI
Record Dates: First submitted 2018-05-17; First posted 2018-06-06 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Colorectal Carcinoma; Soft Tissue Sarcoma
Keywords: Next Generation Sequencing; Exome; RNA sequencing; Soft-tissue sarcoma; Colorectal carcinoma
MeSH Terms: conditions — Colorectal Neoplasms; Sarcoma | interventions — High-Throughput Nucleotide Sequencing; Base Sequence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For each participant, biological specimens will be collected for molecular analysis :
  * Whole blood sample for constitutional characteristics
  * Tumor sample (fresh-frozen or formalin-fixed paraffin embedded)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- STS: Patients with advanced/metastatic soft-tissue sarcoma
  Interventions: Genetic: Next Generation Sequencing (NGS): exome, RNA seq
- CCR: Patients with metastatic colorectal carcinoma
  Interventions: Genetic: Next Generation Sequencing (NGS): exome, RNA seq

INTERVENTIONS:
Genetic: Next Generation Sequencing (NGS): exome, RNA seq — Tumor and blood samples will be sequenced at medium-high coverage at the whole genome (exome) and transcriptome levels (RNA Seq). This will allow detecting variants in a larger set of samples even though only from the main clone will be precisely measured. The whole exome will be performed at a mean coverage of at least 60x for the normal DNA samples and 120x for the tumor DNA samples. The transcriptome of the tumor will be performed at enough depth of coverage to detect gene fusions, transcriptome variants and measure the digital expression of already annotated isoforms.
  For both sequencing configurations:
  * Data from each cancer and normal genome will be analysed for the presence of somatic variants.
  * DNA and RNA sequencing results will be integrated.
  * Technical replication for the mutations / chromosome alterations / transcript fusions that most likely drive the tumour process will be performed via Target Resequencing of the genomic / coding regions of interest.

SUMMARY:
Next Generation Sequencing in cancer: a feasibility study in France to assess sample circuit and to perform analyzes within a limited time.

DETAILED DESCRIPTION:
The first France disease genomic medicine program in the field of cancer has been retained by the 2025 Genomic Medicine France Plan. This program, called MULTIPLI encompasses two innovative personalized medicine clinical trials in soft-tissue sarcoma and colorectal carcinoma involving targeted molecules according to the tumor profile of each patient.

This 1st clinical research program aims implementing exome sequencing and RNA sequencing to determine the genomic profile and to provide a therapeutic decision for each patient. Genomic analyzes will be performed on different technical platforms: samples will be collected in each investigating center, nucleic acids extraction will be performed on two genetic platforms, Inca labeled and identified for the purpose of this study: Institut Bergonié and Hôpital Européen Georges Pompidou. CNRGH (Centre National de Recherche en Génomique Humaine) was retained for operational platform genomics and Institut Bergonie for bioinformatics data processing. Each genomic profile will be discussed within a multidisciplinary tumor board which aims at providing a therapeutic decision for each patient and to propose a targeted treatment in case of actionable molecular alteration.

The purpose of this program is to perform analysis on a set of gene, in order to provide results no more than after 6 weeks after the sample arrival on the biopathological platform. This gene panel analysis is based on the predefined list of genes that are direct targets of the drugs available in the MULTIPLI program.

Before implanting this program in a large-scale launch, it was essential to set up a pilot study in order to evaluate both sample's management between several platforms, and the time to report the results, and to verify that it was in line with the objectives set.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Disease: Advanced and/or metastatic soft-tissue sarcoma OR metastatic carcinoma
* Patient consenting to tumor sequencing, secondary reuse of their data
* Patient informed about this study

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients included in this prospective cohort study are patients who have previously consented to tumor sequencing either as part of others studies or as part of standard care (voluntary signed informed consent). Two participating centers have been retained.
  Samples used (blood and tumor) are issued from these previous collection and analyzed for the same purpose: no additional samples will be collected.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2017-09-21 (Actual); Study Completion 2017-09-21 (Actual)

PRIMARY OUTCOMES:
Delay time to send a validated exome sequencing report from sample receipt | an average of 6 weeks
  The time delay between the date of sample receipt by the platform and the date of dispatch of a validated MTB report to physician

SECONDARY OUTCOMES:
The rate of patients with samples received by Platform for whom a validated exome sequencing report is available | Throughout the study period, on average of 3 months
  Rate of patients for whom a report was transmitted, within the patients for whom the samples were received by the platforms
Delay time to send a validated exome sequencing report from signature to informed consent by the patient | an average of 8 weeks
  The time delay between the date of informed consent signature and the date of dispatch of a validated MTB report to physician
The rate of patients with signed informed consent for whom a validated exome sequencing report is available | Throughout the study period, on average of 3 months
  Rate of patients for whom a report was transmitted, within the patients for whom signed consent has been signed
Delay time to receive sample on Platform from signature of informed consent | on average of 2 weeks
  The time delay between the date of informed consent signature and the date of sample receipt on platform
The rate of patients with signed informed consent for whom samples have been received by platform | Throughout the study period, on average of 3 months
  Rate of patients for whom samples have been received by platform, within the patients for whom signed consent has been signed
Delay time to receipt nucleic acids on CNRGH from samples receipt on platform | on average of 1 week
  The time delay between the date of sample receipt on platform and the date of nucleic acids receipt on CNRGH
The rate of patients with samples sending date completed on electronic case for whom samples have been received by platform | Throughout the study period, on average of 3 months
  Rate of patients for whom samples have been received by platform, within the patients for whom sending date has been completed on electronic case
The rate of patients with samples received on platform for whom these samples have been qualified in first step by platform and nucleic acids have been received by CNRGH | Throughout the study period, on average of 3 months
  Rate of patients for whom samples have been qualified in first step by platform and nucleic acids received by CNRGH, within the patients for whom samples have been received by platform
The rate of patients with samples received on Platform for whom these samples have been qualified in second step by platform and nucleic acids have been received by CNRGH | Throughout the study period, on average of 3 months
  Rate of patients for whom samples have been qualified in second step by platform and nucleic acids received by CNRGH, within the patients for whom samples have been received by platform
The rate of patients with samples received on platform for whom these samples have been qualified in first and second step by Platform and nucleic acids have been received by CNRGH | Throughout the study period, on average of 3 months
  Rate of patients for whom samples have been qualified in first and second step by platform and nucleic acids received by CNRGH, within the patients for whom samples have been received by platform
Delay time to receive all sequencing files from nucleic acids receipt on CNRGH | on average of 3 weeks
  The time delay between the date of nucleic acids receipt on CNRGH and the date of receipt of all sequencing files by bioinformatic platform
The rate of patients with nucleic acids received on CNRGH for whom all sequencing files have been qualified by bioinformatics platform | Throughout the study period, on average of 3 months
  Rate of patients for whom all sequencing files have been qualified by bioinformatics platform, within the patients for whom samples have been received by CNRGH
The rate of patients with nucleic acids received on CNRGH for whom sequencing have been qualified by CNRGH | Throughout the study period, on average of 3 months
  Rate of patients for whom sequencing have been qualified by CNRGH, within the patients for whom samples have been received by CNRGH
Delay time to receive bioinformatics analysis for interpretation from availability of all sequencing files | on average of 1 week
  The time delay between the date of receipt of all sequencing files by bioinformatics platform and the date of receipt of bioinformatics analysis by biologist for interpretation
The rate of patients with sequencing files received by bioinformatic Platform for whom these files have been qualified for analysis | Throughout the study period, on average of 3 months
  Rate of patients for whom all sequencing file have been qualified by bioinformatic platform, within the patients for whom all sequencing file have been received by bioinformatic platform
The rate of patients with sequencing files received by bioinformatic Platform for whom analysis have been transmitted for interpretation | Throughout the study period, on average of 3 months
  Rate of patients for whom bioinformatic analysis have been transmitted for interpretation, within the patients for whom all sequencing file have been received by bioinformatic platform
Delay time to send a validated exome sequencing report from availability of bioinformatic analysis | on average of 1 week
  The time delay between the date of bioinformatic analysis availability for interpretation and the date of dispatch of a validated MTB report to physician
The rate of patients with bioinformatic analysis available for interpretation for whom biological interpretation has been performed | Throughout the study period, on average of 3 months
  Rate of patients for whom bioinformatic analysis has been interpreted by biologist, within the patients for whom bioinformatics analysis have been transmitted
The rate of patients with bioinformatic analysis available for interpretation for whom results has been discussed by MTB | Throughout the study period, on average of 3 months
  Rate of patients for whom biological report has been discussed by MTB, within the patients for whom bioinformatics analysis have been transmitted

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Institut Bergonié, Bordeaux
  - CEA / Centre National de Recherche en Génomique Humaine, Évry
  - Hôpital Européen Georges Pompidou, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] FGM 2025 Workflow Study Group (Alliance nationale des Sciences de la Vie et de la Sante); Auzanneau C, Bacq D, Bellera C, Blons H, Boland A, Boucheix M, Bourdon A, Chollet E, Chomienne C, Deleuze JF, Delmas C, Dinart D, Esperou H, Geillon F, Geneste D, Italiano A, Jean D, Khalifa E, Laizet Y, Laurent-Puig P, Lethimonnier F, Levy-Marchal C, Lucchesi C, Malle C, Mancini P, Mathoulin-Pelissier S, Meyer V, Marie-Ange P, Perkins G, Sellan-Albert S, Soubeyran I, Wallet C. Feasibility of high-throughput sequencing in clinical routine cancer care: lessons from the cancer pilot project of the France Genomic Medicine 2025 plan. ESMO Open. 2020 Jul;5(4):e000744. doi: 10.1136/esmoopen-2020-000744. PMID 32713836